CLINICAL TRIAL: NCT05262205
Title: Bispectral Index Monitoring In Pediatric Cataract Surgery: A Comparative Study Using Propofol- Midazolam Versus Sevoflurane Anesthesia
Brief Title: Bispectral Index Monitoring In Pediatric Cataract Surgery: A Comparative Study Using Propofol-Midazolam Versus Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Zahraa Ibrahim Zamzm, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD.21.03.449.R1-2021/04/2021
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Ophthalmic
Keywords: propofol; ocular alignment; TIVA

STUDY DESIGN:
Intervention Model Description: 2 groups, each is 50 child randomly allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sevoflurane group with BIS monitor for depth of anesthesia (Active Comparator): child will be anesthetized with sevoflurane 2% and atracurium 0.25mg/kg and paracetamol 15mg/kg, then bispectral index will be recorded after intubation and every five minutes till end of surgery. Position of the globe will recorded every five minutes. Angle of deviation of the globe will be calculated via withdrawing horizontal line passing from the lateral and medial canthi, and another vertical one passing the medial canthus(90-0--90 degree). Bis should be 40-65 to ensure adequate depth of anesthesia. If more than 65 or less than 40, sevoflurane concentration will be adjusted till having the target range. pupillary dilation in surgical eye will be assessed after speculum insertion, 20 minutes after speculum insertion, and before speculum removal by pupil ruler((pupil gauge), whether it will be maintained or not (considered maintained if pupil size equal or more than 5mm).
  Interventions: Other: measuring depth of anesthesia and its relation to the globe
- propofol-midazolam group with BIS monitor for depth of anesthesia (Active Comparator): Child will be anesthetized with midazolam 0.05 mg/kg IV bolus and propofol 1mg/kg IV bolus, paracetamol 15mg\kg IV infusion, and atracurium 0.25mg/kg IV bolus ,then anesthesia will be maintained with propofol infusion according to Mcfarlan protocol, then BIS will be recorded after intubation and every five minutes till end of surgery. Position of the globe will recorded every five minutes till the end of surgery. Angle of deviation will be calculated in same way as group A. Bis should be 40-65. If more than 65 or less than 40, sevoflurane concentration will be adjusted till having the target range. pupillary dilation in surgical eye will be assessed after speculum insertion, 20 minutes after speculum insertion, and before speculum removal by pupil ruler((pupil gauge) and will be observed all over the surgery with the help of surgeon feedback whether it will be maintained or not (considered maintained if pupil size equal or more than 5mm).
  Interventions: Other: measuring depth of anesthesia and its relation to the globe

INTERVENTIONS:
Other: measuring depth of anesthesia and its relation to the globe — measuring feasibility of BIS monitor in detecting depth of anesthesia in pediatric population and whether it will be beneficial as a tool for helping anesthesiologist in maintaining central globe alignment

SUMMARY:
Ocular alignment will be studied in children having cataract surgery that will be divided into two groups, one group will be anesthetized using sevoflurane anesthesia (group A), and the other will be anesthetized by midazolam bolus and propofol infusion (total intravenous anesthesia, TIVA) (group B). in both groups depth of anesthesia will be monitored by bispectral index monitor.

DETAILED DESCRIPTION:
After signing the informed consent by children parent, child will be transferred to the operating room and will be connected to pulse oximetry, non invasive blood pressure and electrocardiogram(ECG), child will be anesthetized by sevoflurane 8% for cannula insertion, then in Group A, sevoflurane will be continued with 2%, and iv atracurium 0.25mg/kg, and paracetamol 15mg/kg iv will be given. In group B, sevoflurane will be discontinued and propofol bolus1mg/kg iv, midazolam 0.05 mg/kg iv, atracurium 0.25 iv, and paracetamol 15mg/kg iv then propofol infusion will start immediately according to McFarlan protocol for manual syringe pump for pediatrics. For first 10 minutes 15mg/kg, second 10 minutes 13mg/kg, third 10 minutes 13mg/kg, fourth 10 minutes 11mg/kg, fifth 10 minutes 11mg/kg, and will be continued on this rate for the end of surgery. Bispectral index monitor(Covidien, Germany) will be attached to child forehead after cleansing it with alcohol 70%. after adequate jaw relaxation , trachea will be intubated with adequate size endotracheal tube and attached to anesthesia machine ( General electric, Carestation 650).Volume controlled ventilation (VCV) will start with tidal volume(VT) 6-8 ml/kg, respiratory rate (RR)16-20 according to end-tidal carbon dioxide (CO2)35-40mmhg. Flow of fresh gas rate 2 l/minute. standard circuit system connection for pediatric will be used. Heart rate ,peripheral oxygen saturation (SPO2), non invasive blood pressure, end-tidal carbon dioxide (ETCO2), and bispectral index monitor will be measured every 5 minutes. 6 ml/kg of ringer will be given infusion slowly.

ELIGIBILITY:
Inclusion Criteria:

0-children American society of anesthesiologist (ASA )grade l, ll of both sex 0-congenital or traumatic cataract

Exclusion Criteria:

0- syndromes involving cataract. 0- children with neurologic disorders. 0- children on anti-psychotic medication. 0- hypersensitivity to any anesthetic used.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
assessing depth of anesthesia and its relation to ocular alignment | after intubation and every five minutes till end of surgery
  depth of anesthesia will be measured using bispectral index monitor (BIS) monitor and position of the globe will be assessed and related to it by measuring the angle of deviation in degrees. Then, correlation the findings using pearson correlation co-effecient

SECONDARY OUTCOMES:
pupillary dilatation | after insertion of the speculum by 10 minutes and 20 minutes
  pupil of surgical eye is dilated with phenylephrine 2.5%. assessing wether pupillary dilatation will be maintained during anesthesia (> or aqual to 5 mm) or not by using pupil gauge.

OTHER OUTCOMES:
post emergence agitation | after extubation and for 30 minutes later.
  the child will be assessed with Watcha scale. If score is 4 he is considered agitated

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Abd-Elmagid, professor, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCann ME, Bacsik J, Davidson A, Auble S, Sullivan L, Laussen P. The correlation of bispectral index with endtidal sevoflurane concentration and haemodynamic parameters in preschoolers. Paediatr Anaesth. 2002 Jul;12(6):519-25. doi: 10.1046/j.1460-9592.2002.00886.x. PMID 12139593
- [Background] Johar SR, Savalia NK, Vasavada AR, Gupta PD. Epidemiology based etiological study of pediatric cataract in western India. Indian J Med Sci. 2004 Mar;58(3):115-21. PMID 15051906
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Darlong V, Garg R, Pandey R, Khokhar S, Chandralekha, Sinha R, Punj J, Sinha R. Evaluation of minimal dose of atracurium for cataract surgery in children: A prospective randomized double-blind study. Saudi J Anaesth. 2015 Jul-Sep;9(3):283-8. doi: 10.4103/1658-354X.154711. PMID 26240547
- [Background] Degoute CS, Macabeo C, Dubreuil C, Duclaux R, Banssillon V. EEG bispectral index and hypnotic component of anaesthesia induced by sevoflurane: comparison between children and adults. Br J Anaesth. 2001 Feb;86(2):209-12. doi: 10.1093/bja/86.2.209. PMID 11573661
- [Background] Gilbert C, Foster A. Childhood blindness in the context of VISION 2020--the right to sight. Bull World Health Organ. 2001;79(3):227-32. Epub 2003 Jul 7. PMID 11285667
- [Background] Kook KH, Chung SA, Park S, Kim DH. Use of the Bispectral Index to Predict Eye Position of Children during General Anesthesia. Korean J Ophthalmol. 2018 Jun;32(3):234-240. doi: 10.3341/kjo.2017.0104. Epub 2018 May 15. PMID 29770643
- [Background] Pieters BJ, Penn E, Nicklaus P, Bruegger D, Mehta B, Weatherly R. Emergence delirium and postoperative pain in children undergoing adenotonsillectomy: a comparison of propofol vs sevoflurane anesthesia. Paediatr Anaesth. 2010 Oct;20(10):944-50. doi: 10.1111/j.1460-9592.2010.03394.x. Epub 2010 Aug 24. PMID 20735801
- [Background] Rodgers A, Cox RG. Anesthetic management for pediatric strabismus surgery: Continuing professional development. Can J Anaesth. 2010 Jun;57(6):602-17. doi: 10.1007/s12630-010-9300-x. PMID 20393822
- [Background] Rossiter JD, Wood M, Lockwood A, Lewis K. Operating conditions for ocular surgery under general anaesthesia: an eccentric problem. Eye (Lond). 2006 Jan;20(1):55-8. doi: 10.1038/sj.eye.6701789. PMID 15650757
- [Background] Bajwa SA, Costi D, Cyna AM. A comparison of emergence delirium scales following general anesthesia in children. Paediatr Anaesth. 2010 Aug;20(8):704-11. doi: 10.1111/j.1460-9592.2010.03328.x. PMID 20497353
- [Background] Fodale V, Pratico C, Santamaria LB. Coadministration of propofol and midazolam decreases bispectral index value as a result of synergic muscle relaxant action on the motor system. Anesthesiology. 2004 Sep;101(3):799; author reply 800-1. doi: 10.1097/00000542-200409000-00033. No abstract available. PMID 15329609
- [Background] Anderson BJ, Bagshaw O. Practicalities of Total Intravenous Anesthesia and Target-controlled Infusion in Children. Anesthesiology. 2019 Jul;131(1):164-185. doi: 10.1097/ALN.0000000000002657. PMID 30920966
- Available data/document: Study Protocol — http://irb.mans.edu.eg